CLINICAL TRIAL: NCT00733499
Title: A Prospective, Randomised, Single Blinded Study Comparing the Pain, Biological Fixation and Outcomes of Patients With LCS Complete Duofix or LCS Porocoat Knee Systems
Brief Title: A Study to Determine the Difference in Low Contact Stress (LCS) Duofix Versus Low LCS Porocoat Knee Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT 05/28
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty, replacement, Knee, LCS Duofix, Porocoat
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCS Complete Duofix (Other): 102 patients
  Interventions: Device: LCS Complete Duofix
- LCS Complete Porocoat (Active Comparator): 104 patients
  Interventions: Device: LCS Complete Porocoat

INTERVENTIONS:
Device: LCS Complete Duofix — Orthopaedic implant for total knee replacement with Duofix biological fixation surfaces
  Arms: LCS Complete Duofix
Device: LCS Complete Porocoat — Orthopaedic implant for total knee replacement with Porocoat biological fixation surfaces
  Arms: LCS Complete Porocoat

SUMMARY:
The primary objective of this investigation is to test the hypothesis that the Duofix Tibial component results in a reduction of immediate postoperative pain compared to the LCS Porocoat version.

DETAILED DESCRIPTION:
The secondary objectives of this investigation are to evaluate the clinical and patient outcomes, biological fixation and survivorship associated with the LCS Duofix and Porocoat knee system over 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects who present with idiopathic osteoarthritis, rheumatoid arthritis, post traumatic arthritis or any other pathology that in the opinion of the clinical investigator requires a primary total knee arthroplasty and who are considered suitable for treatment with a cementless mobile bearing knee system (LCS Complete).
* Subjects who in the opinion of the Clinical Investigator are considered to be suitable for treatment with both the investigational devices, according to the indications specified in the package insert leaflet.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
* Subjects with a known history of poor compliance to medical treatment.
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects involved in Medical-Legal claims.
* Subjects who have participated in a clinical study with an investigational product in the last month.
* Subjects who are currently involved in any injury litigation claims.
* Revision of an existing knee implant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2009-10-01 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Musgrave Park Hospital, Belfast, Ireland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was operated on 26 September 2006 and recruitment lasted for 28 months with the last patient operated on 20th January 2009.
Pre-assignment Details: Consent was taken for 232 knees. 10 subjects were deemed unfit for surgery, 5 subjects were deemed ineligible for the study and 12 subjects were not randomised for the study. This left 205 subjects in the safety population that could be randomised for the study.
Groups:
- LCS Complete Duofix: LCS Complete Duofix patients : Orthopaedic implant for total knee replacement with Duofix biological fixation surfaces
- LCS Complete Porocoat: LCS Complete Porocoat patients : Orthopaedic implant for total knee replacement with Porocoat biological fixation surfaces
Period: Pre-operative
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Started | 102 | 103 (A death occurred prior to surgery which left a total of 102 participants)
Completed | 102 | 102
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: 3 Months Follow-up
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Started | 102 | 102
Completed | 101 | 100
Not Completed | 1 | 2
Not completed — Death | 1 | 2
Period: 6 Months Follow-up
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Started | 101 | 100
Completed | 101 | 97
Not Completed | 0 | 3
Not completed — Death | 0 | 2
Not completed — Adverse Event | 0 | 1
Period: 12 Months Follow-up
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Started | 101 | 97
Completed | 99 | 96
Not Completed | 2 | 1
Not completed — Death | 2 | 1
Period: 24 Months Follow-up
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Started | 99 | 96
Completed | 99 | 95
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: 5 Year Followup
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Started | 91 | 78
Completed | 70 | 53
Not Completed | 21 | 25
Not completed — Adverse Event | 2 | 2
Not completed — Non device related AE | 0 | 1
Not completed — Revision of Study Implant | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 13 | 19
Not completed — missing, unable to locate | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1
Period: 10 Year Followup
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Started | 46 | 32
Completed | 26 | 13
Not Completed | 20 | 19
Not completed — Death | 9 | 7
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 5 | 5
Not completed — missing, unable to locate | 0 | 2

BASELINE CHARACTERISTICS:
Population: The number of participants in the intent to treat population (All eligible subjects, admitted to the study that receive the allocated treatment, and have at least one usable post-treatment assessment).
Groups:
- Total: Total of all reporting groups
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.39 (8.98) | 70.49 (8.97) | 70.94 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 62 | 134
  Male | 30 | 40 | 70
Region of Enrollment [Count of Participants; unit: Participants]
  Ireland: Ireland | 102 | 102 | 204

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Mean VAS Pain Score Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 12 Months.
Description: The visual analog scale (VAS) pain score asks the subject to place a vertical mark anywhere on a horizontal line (that is approximately 10 cm long) with 'No pain' listed on the left (scored as 0) and 'Very severe pain' labeled on the right (scored as 10). The subject is instructed to indicate the amount of pain they feel in their knee joint
Time Frame: 12 Months Post Surgery
Population: The number of participants analysed is based on the number of case report forms measuring the VAS pain score that we have in our database at the 12 month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 87 | 87
units on a scale | 2.51 (2.226) | 2.53 (2.166)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.9478, t-test, 2 sided

2. Secondary Outcome: Comparative Evaluation of Any Variability in Functional Recovery Using the Oxford Knee Score Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at Pre-op.
Description: The Oxford Knee Score questionnaire consists of 12 questions each with a choice of responses and is designed to evaluate the subjects' perception of the condition and functionality of their affected joint and the impact that it has on their normal daily activities. Overall scores range from 0 (most severe symptoms) to 48 (least symptoms) with 48 being the best outcome.
Time Frame: Pre-op
Population: The number of participants analysed is based on the number of case report forms measuring the Oxford Knee Score that we have in our database at the preop time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 102 | 102
units on a scale | 45.81 (4.393) | 45.40 (5.357)
Statistical Analysis 1: Comparison: LCS Complete Duofix; Test type: Other; p = 0.5490, t-test, 2 sided

3. Secondary Outcome: Comparative Evaluation of Any Variability in Functional Recovery Using the Oxford Knee Score Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 3 Months.
Description: as for outcome 2
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 96 | 92
units on a scale | 28.66 (8.993) | 29.45 (8.224)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.5312, t-test, 2 sided

4. Secondary Outcome: Comparative Evaluation of Any Variability in Functional Recovery Using the Oxford Knee Score Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 6 Months.
Description: as for outcome 2
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 87 | 87
units on a scale | 25.16 (6.963) | 26.10 (6.429)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.3549, t-test, 2 sided

5. Secondary Outcome: Comparative Evaluation of Any Variability in Functional Recovery Using the Oxford Knee Score Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 12 Months.
Description: as for outcome 2
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 97 | 93
units on a scale | 24.70 (8.341) | 27.17 (9.022)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.0513, t-test, 2 sided

6. Secondary Outcome: Comparative Evaluation of Any Variability in Functional Recovery Using the Oxford Knee Score Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 24 Months.
Description: as for outcome 2
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 99 | 94
units on a scale | 23.39 (7.783) | 25.68 (9.172)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.0629, t-test, 2 sided

7. Secondary Outcome: Comparative Evaluation of Any Variability in Functional Recovery Using the Oxford Knee Score Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 60 Months.
Description: as for outcome 2
Time Frame: 60 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 80 | 75
units on a scale | 24.05 (8.322) | 27.25 (10.145)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.0327, t-test, 2 sided

8. Secondary Outcome: Comparative Evaluation of Any Variability in Functional Recovery Using the Oxford Knee Score Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 120 Months.
Description: as for outcome 2
Time Frame: 120 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 49 | 37
units on a scale | 22.04 (7.514) | 25.49 (10.197)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.0883, t-test, 2 sided

9. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Mental Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at Pre-op.
Description: The SF-12 consists of 12 questions that explores issues that apply to people have many different types of treatment, and in all different states of health, from good to bad. The mental composite score ranges from 0 to 100, where 0 indicates the lowest level of health and 100 indicates the highest level of health.
Time Frame: pre-op
Population: The number of participants analysed is based on the number of case report forms measuring the SF-12 that we have in our database at the preop time point. Please note-due to a discrepancy in an early version of the SF12 case report from, a complete score could not be calculated which reflected in missing counts for early visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 13 | 16
units on a scale | 47.39 (9.464) | 47.54 (8.084)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.6801, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Mental Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 3 Months.
Description: as for outcome 9
Time Frame: 3 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 38 | 34
units on a scale | 49.87 (9.931) | 48.21 (9.784)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.4779, t-test, 2 sided

11. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Mental Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 6 Months.
Description: as for outcome 9
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 39 | 35
units on a scale | 52.54 (9.532) | 51.99 (9.261)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.8007, t-test, 2 sided

12. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Mental Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 12 Months.
Description: as for outcome 9
Time Frame: 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 66 | 67
units on a scale | 51.60 (10.905) | 49.83 (10.022)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.3317, t-test, 2 sided

13. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Mental Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 24 Months.
Description: as for outcome 9
Time Frame: 24 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 78 | 79
units on a scale | 52.88 (8.597) | 52.81 (8.662)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.8955, t-test, 2 sided

14. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Mental Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 60 Months.
Description: as for outcome 9
Time Frame: 60 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 72 | 65
units on a scale | 49.87 (11.395) | 47.38 (11.757)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.2116, t-test, 2 sided

15. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Mental Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 120 Months.
Description: as for outcome 9
Time Frame: 120 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 49 | 37
units on a scale | 54.85 (7.877) | 53.49 (9.821)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.4776, t-test, 2 sided

16. Secondary Outcome: Survivorship Analysis
Description: The survival of each group is assessed using Kaplan-Meier curves. Revision for any reason constitutes an event.
Time Frame: 5 Years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 90 | 81
Percentage of Participants | 100 [100.0 to 100.0] | 98.9 [92.1 to 99.8]

17. Secondary Outcome: Survivorship Analysis
Description: The survival of each group is assessed using Kaplan-Meier curves. Revision for any reason constitutes an event.
Time Frame: 9.99 years
Population: 10 Year survivorship could not be calculated due to N <40 but could be calculated at 9.99 years.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 38 | 34
Percentage of Participants | 100 [100.0 to 100.0] | 98.9 [92.1 to 99.8]
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.2935, t-test, 2 sided

18. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Physical Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at Preop.
Description: The SF-12 consists of 12 questions that explores issues that apply to people have many different types of treatment, and in all different states of health, from good to bad. The physical composite score ranges from 0 to 100, where 0 indicates the lowest level of health and 100 indicates the highest level of health.
Time Frame: preop
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 13 | 16
units on a scale | 30.8 (6.085) | 24.81 (3.089)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.0062, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Physical Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 3 Months.
Description: as for outcome 18
Time Frame: 3 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 38 | 34
units on a scale | 35.50 (8.927) | 34.64 (9.171)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.6896, t-test, 2 sided

20. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Physical Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 6 Months.
Description: as for outcome 18
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 39 | 35
units on a scale | 36.58 (8.411) | 33.31 (8.800)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.1076, t-test, 2 sided

21. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Physical Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 12 Months.
Description: as for outcome 18
Time Frame: 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 66 | 67
units on a scale | 36.76 (9.353) | 36.56 (9.346)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.9042, t-test, 2 sided

22. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Physical Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 24 Months.
Description: as for outcome 18
Time Frame: 24 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 78 | 79
units on a scale | 37.41 (10.577) | 37.49 (9.693)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.9637, t-test, 2 sided

23. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Physical Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 60 Months.
Description: as for outcome 18
Time Frame: 60 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 72 | 65
units on a scale | 36.52 (10.802) | 32.93 (10.259)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.0485, t-test, 2 sided

24. Secondary Outcome: Comparative Evaluation of Any Variability in Quality of Life Assessed by SF-12 (Physical Composite) Questionnaire Between Subjects Receiving LCS Complete Duofix™ and Porocoat® Knee Systems at 120 Months.
Description: as for outcome 18
Time Frame: 120 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 49 | 37
units on a scale | 40.73 (10.465) | 40.78 (10.701)
Statistical Analysis 1: Comparison: LCS Complete Duofix vs LCS Complete Porocoat; Test type: Other; p = 0.9813, t-test, 2 sided

25. Secondary Outcome: Number of Participants With Tibial Radiolucency, 0-1mm
Description: Zonal Analysis of the 6 zones of the tibial component was determined from the post operative radiographs. Osteo-fixation was graded using the following system 0-1 mm radiolucencies will be classed as fixated, 1-2mm not fixated, >2mm unstable.
Time Frame: 3 months to 120 months
Population: Subjects within safety population with complete, available data.
Measure: Count of Participants; unit: Participants
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 102 | 102
Participants
  3 months: number analyzed (Participants) | 92 | 75
  3 months | 13 | 20
  12 months: number analyzed (Participants) | 90 | 84
  12 months | 14 | 27
  60 months: number analyzed (Participants) | 73 | 74
  60 months | 14 | 18
  120 months: number analyzed (Participants) | 37 | 30
  120 months | 6 | 10

26. Secondary Outcome: Number of Participants With Tibial Radiolucency, 1mm-2mm
Description: as for outcome 25
Time Frame: 3 months to 120 months
Population: Subjects within safety population with complete, available data.
Measure: Count of Participants; unit: Participants
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 102 | 102
Participants
  3 months: number analyzed (Participants) | 92 | 75
  3 months | 13 | 20
  12 months: number analyzed (Participants) | 90 | 84
  12 months | 14 | 31
  60 months: number analyzed (Participants) | 73 | 74
  60 months | 21 | 32
  120 months: number analyzed (Participants) | 37 | 30
  120 months | 6 | 8

27. Secondary Outcome: Number of Participants With Tibial Radiolucency, Greater Than 2mm
Description: as for outcome 25
Time Frame: 3 months to 120 months
Population: Subjects within safety population with complete, available data.
Measure: Count of Participants; unit: Participants
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
Number analyzed (Participants) | 102 | 102
Participants
  3 months: number analyzed (Participants) | 92 | 75
  3 months | 3 | 6
  12 months: number analyzed (Participants) | 90 | 84
  12 months | 3 | 5
  60 months: number analyzed (Participants) | 73 | 74
  60 months | 5 | 6
  120 months: number analyzed (Participants) | 37 | 30
  120 months | 1 | 1

ADVERSE EVENTS:
Time Frame: All participants had reached the 10 year follow-up visit at the time of uploading adverse events
Description: Final assessment of adverse events were classified by organ system class in lieu of specific adverse event terms.
Arm/Group | LCS Complete Duofix | LCS Complete Porocoat
All-Cause Mortality (participants affected / at risk) | 27/102 | 33/103
Serious Adverse Events (participants affected / at risk) | 58/102 | 68/103
Other Adverse Events (participants affected / at risk) | 17/102 | 17/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCS Complete Duofix (N=102) | LCS Complete Porocoat (N=103)
Cardiac Disorder (Cardiac disorders) | 5 (6) | 8 (9)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 2 (4)
Infections and infestations (Infections and infestations) | 10 (12) | 9 (11)
General disorders and administration site conditions (General disorders) | 5 (6) | 6 (6)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 7 (14) | 10 (18)
Investigations (Investigations) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 23 (34) | 27 (34)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (13) | 9 (12)
Nervous System disorders (Nervous system disorders) | 7 (7) | 10 (11)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCS Complete Duofix (N=102) | LCS Complete Porocoat (N=103)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 17 (50) | 17 (61) — Reported as AEs and not SAEs. Final assessment of adverse events were classified by organ system class in lieu of specific adverse event terms.

LIMITATIONS AND CAVEATS:
This is a single surgeon/site study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
DePuy reserves the right to review the contents of publications in advance.The PI may freely disclose the trial results only after DePuy has been given the opportunity of reviewing the proposed results communications at least 30 days prior to the intended release.DePuy will advise the PI of any perceived errors,omissions or corrections but the PI will retain final editorial control.In case of disagreement,DePuy and the PI will make every effort to meet in order to discuss and resolve any issues.